CLINICAL TRIAL: NCT04749368
Title: A Phase 2 Multicenter, Randomized, Open-label Study to Investigate the Safety and Efficacy of BRII-835 (VIR-2218) and BRII-179 (VBI-2601) Combination Therapy for the Treatment of Chronic Hepatitis B Virus (HBV) Infection
Brief Title: Study to Investigate the Safety and Efficacy of BRII-835 and BRII-179 Combination Therapy Treating Chronic Hepatitis B Virus (HBV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brii Biosciences Limited (Industry)
Collaborators: Vir Biotechnology, Inc. (Industry); VBI Vaccines Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRII-179-835-001
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B Virus; Chronic Hepatitis B; HBV; Hepatitis
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort A (Experimental): Participants will receive BRII-835 (VIR-2218) for 32 weeks
  Interventions: Drug: BRII-835 (VIR-2218)
- Cohort B (Experimental): Participants will receive BRII-835 (VIR-2218) and BRII-179 (VBI-2601) with IFN-α up to Week 40
  Interventions: Drug: BRII-835 (VIR-2218); Biological: BRII-179 (VBI-2601) with IFN-α
- Cohort C (Experimental): Participant will receive BRII-835 (VIR-2218) and BRII-179 (VBI-2601) up to Week 40
  Interventions: Drug: BRII-835 (VIR-2218); Biological: BRII-179 (VBI-2601)

INTERVENTIONS:
Drug: BRII-835 (VIR-2218) — BRII-835 (VIR-2218) will be given by subcutaneous injection
Biological: BRII-179 (VBI-2601) with IFN-α — BRII-179 (VBI-2601) with IFN-α will be co-administered by intramuscular injection
  Arms: Cohort B
Biological: BRII-179 (VBI-2601) — BRII-179 (VBI-2601) will be administered by intramuscular injection
  Arms: Cohort C

SUMMARY:
This is an open label, randomized, parallel-group study to evaluate the safety and efficacy of combination treatment BRII-835 (VIR-2218) and BRII-179 (VBI-2601) in adult participants with chronic HBV infection

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 - 60
* Body mass index ≥ 18 kg/m^2 and ≤ 32 kg/m^2
* Chronic HBV infection as defined by a positive serum HBsAg for ≥ 6 months

Exclusion Criteria:

* Any clinically significant chronic or acute medical condition that makes the volunteer unsuitable for participation
* Significant fibrosis or cirrhosis
* History or evidence of drug or alcohol abuse
* History of intolerance to SC or IM injection
* History of chronic liver disease from any cause other than chronic HBV infection
* History of hepatic decompensation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with sustained HBsAg loss during the 48-week follow-up period after NrtI withdrawal | up to Week 96
Number of participants with Adverse Events (AE) | up to Week 96
Number of participants with Serious Adverse Events (SAE) | up to Week 96
Number of participants with abnormalities in clinical laboratory tests | up to Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofei Chen, Study Director — Brii Biosciences Limited
Locations (28):
- Australia (3):
  - Investigative Site 61002, Kingswood, New South Wales
  - Investigative Site 61001, Westmead, New South Wales
  - Investigative Site 61004, Herston, Queensland
- China (9):
  - Investigative Site 88602, Changhua, Taiwan
  - Investigative Site 85201, Hong Kong
  - Investigative Site 85202, Hong Kong
  - Investigative Site 85203, Hong Kong
  - Investigative Site 88601, Kaohsiung, Taiwan
  - Investigative Site 88604, Kaohsiung, Taiwan
  - Investigative Site 85204, NEW Territories, Hong Kong
  - Investigative Site 88603, Taichung, Taiwan
  - Investigative Site 88605, Taipei CITY
- New Zealand (2):
  - Investigative Site 64002, Dunedin Central, Dunedin
  - Investigative Site 64001, Auckland
- Singapore (2):
  - Investigative Site 65001, Singapore
  - Investigative Site 65002, Singapore
- South Korea (5):
  - Investigative Site 82004, Busan
  - Investigative Site 82003, Seongnam-si, Gyeonggi-do
  - Investigative Site 82001, Seoul
  - Investigative Site 82005, Seoul
  - Investigative Site 82002, Seoul
- Thailand (7):
  - Investigative Site 66001, Bangkok
  - Investigative Site 66003, Chiang Mai
  - Investigative Site 66002, Khon Kaen
  - Investigative Site 66005, Nonthaburi
  - Investigative Site 66006, Nonthaburi
  - Investigative Site 66004, Pathum Thani
  - Investigative Site 66007, Songkhla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji Y, Le Bert N, Lai-Hung Wong G, Douglas MW, Lee A, Zhu C, Wang B, Lv J, Li D, Tan Y, Ma H, Chen J, Chen X, Zhu Q, Yuen MF, Bertoletti A. The Impact of Hepatitis B Surface Antigen Reduction via Small Interfering RNA Treatment on Natural and Vaccine (BRII-179)-Induced Hepatitis B Virus-Specific Humoral and Cellular Immune Responses. Gastroenterology. 2025 Jul;169(1):136-149. doi: 10.1053/j.gastro.2025.02.016. Epub 2025 Mar 3. PMID 40043858